CLINICAL TRIAL: NCT00293540
Title: Phase III Randomized Study of Luteal Phase vs. Follicular Phase Surgical Oophorectomy and Tamoxifen in Premenopausal Women With Metastatic Hormone Receptor-Positive Breast Cancer
Brief Title: Luteal vs Follicular Surgical Oophorectomy and Tamoxifen in Premenopausal Women With Metastatic Hormone Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Breast Cancer Research Foundation (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Richard R. Love, Scientific director, International Breast Cancer Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0476
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: metastatic; secondary; Hormone Receptor-Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Ovariectomy; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Surgical oophorectomy in history-estimated mid-luteal phase of menstrual cycle plus Tamoxifen
  Interventions: Procedure: oophorectomy; Drug: Tamoxifen
- B (Active Comparator): Surgical oophorectomy in history-estimated mid-follicular phase of menstrual cycle plus Tamoxifen
  Interventions: Procedure: oophorectomy; Drug: Tamoxifen

INTERVENTIONS:
Procedure: oophorectomy — Excision of an ovary
Drug: Tamoxifen — 20 mg orally every day
  Other Names: Nolvadex

SUMMARY:
This study will determine if hormone receptor positive premenopausal metastatic breast cancer patients who undergo removal of the ovaries in mid-luteal versus mid-follicular phase have a longer survival.

DETAILED DESCRIPTION:
Rationale: Previous research suggests that women who have their ovaries removed as part of their treatment for breast cancer may live longer if the ovarian surgery is performed during the luteal phase (last 14 days of the menstrual cycle) rather than the follicular phase (the first 14 days of the menstrual cycle). The current study will evaluate this important research question in premenopausal women with metastatic hormone receptor-positive breast cancer who will be treated with surgery and tamoxifen.

Purpose: The purpose of this research is to find out if premenopausal women with breast cancer that has spread to other parts of the body live longer if their ovaries are removed during the second half of the menstrual cycle. This study will compare how long women live if they have their ovaries removed during the first half of their menstrual cycle (follicular phase) to how long women live if they have their ovaries removed during the second half of their menstrual cycle (luteal phase). Tamoxifen will also be given to study participants.

Treatment: Study participants will have tests performed in advance of surgery to remove their ovaries. Surgery will be performed within four weeks of these tests. The exact day will be determined by the study participant's menstrual history and by a process called randomization, which is a random decision making process to determine if each study participant will have their surgery during the first or second half of their menstrual cycle. On the day of surgery, blood will be taken immediately prior to surgery and three hours after surgery for hormone tests. After the surgery, study participants will be given tamoxifen in oral pills for daily consumption. Study participants will be asked to return to the hospital every two months for tests and distribution of additional tamoxifen tablets. Treatments will be discontinued for disease progression or unacceptable adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Estrogen receptor or progesterone receptor positive breast cancer
* Premenopausal with regular menstrual cycles

Exclusion Criteria:

* Current oral contraceptives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2006-02; Primary Completion 2014-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Love, MD, Principal Investigator — Ohio State University
Locations (21):
- Ohio State University, Columbus, Ohio, United States
- Dhaka Medical College Hospital, Dhaka, Bangladesh
- China (8):
  - 4th Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Beijing Hospital, Beijing
  - Cancer Institute, Beijing
  - Choa Yang Capital Institute, Beijing
  - National Railroad, Beijing
  - Peoples Hospital, Beijing
  - Qilu Hospital, Jinan
  - Fudan University, Shanghai
- Nizam's Institute, Hyderabaad, India
- Dr. Ciptomanounkusumo General Hospital, Jakarta, Indonesia
- UN. Mayala, Kuala Lumpur, Malaysia
- National Institute of Oncology, Rabat, Morocco
- University College Hospital, Ibadan, Nigeria
- Philippines (5):
  - East Avenue Medical Center, Manila
  - Jose Reyes, Manila
  - Philippines General Hospital, Manila
  - Rizal, Manila
  - Vicente Sotto Hospital, Manila
- Hospital K, Hanoi, Vietnam

REFERENCES:
- [Derived] Love RR, Hossain SM, Hussain MM, Mostafa MG, Laudico AV, Siguan SS, Adebamowo C, Sun JZ, Fei F, Shao ZM, Liu Y, Akram Hussain SM, Zhang B, Cheng L, Panigaro S, Walta F, Chuan JH, Mirasol-Lumague MR, Yip CH, Navarro NS Jr, Huang CS, Lu YS, Ferdousy T, Salim R, Akhter C, Nahar S, Uy G, Young GS, Hade EM, Jarjoura D. Luteal versus follicular phase surgical oophorectomy plus tamoxifen in premenopausal women with metastatic hormone receptor-positive breast cancer. Eur J Cancer. 2016 Jun;60:107-16. doi: 10.1016/j.ejca.2016.03.011. Epub 2016 Apr 20. PMID 27107325

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A Mid-luteal Surgery | B Mid-follicular Surgery
Started | 122 | 127
Completed | 115 | 119
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Mid-luteal Surgery | B Mid-follicular Surgery | Total
Number analyzed (Participants) | 115 | 119 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (5.4) | 38.6 (5.7) | 38.8 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 119 | 234
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 1 | 0 | 1
  Bangladesh | 50 | 48 | 98
  Morocco | 0 | 1 | 1
  Philippines | 28 | 26 | 54
  China | 21 | 27 | 48
  Malaysia | 3 | 3 | 6
  Nigeria | 6 | 6 | 12
  Indonesia | 3 | 4 | 7
  Taiwan | 3 | 4 | 7
Dominant metastatic site [Number; unit: participants]
  Soft tissue | 76 | 83 | 159
  Bone | 20 | 25 | 45
  Viscera | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Assess whether patients who undergo surgical oophorectomy in the history-estimated mid-luteal phase of their menstrual cycles survive longer than patients who undergo this surgery in the history-estimated mid-follicular phase of their menstrual cycles.
Time Frame: Up to 9 years
Population: Analyzed all patients with followup data
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | A Mid-luteal Surgery | B Mid-follicular Surgery
Number analyzed (Participants) | 115 | 119
years | 2.14 [1.53 to 2.67] | 2.00 [1.61 to 2.31]

ADVERSE EVENTS:
Arm/Group | A Mid-luteal Surgery | B Mid-follicular Surgery
Serious Adverse Events (participants affected / at risk) | 0/115 | 1/119
Other Adverse Events (participants affected / at risk) | 0/115 | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Mid-luteal Surgery (N=115) | B Mid-follicular Surgery (N=119)
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Pt developed deep vein thrombosis and was successfully treated with anti-coagulants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes